CLINICAL TRIAL: NCT02917720
Title: Multicenter Prospective Trial After 1st or 2nd Unsuccessful Treatment Discontinuation in Chronic Myeloid Leukemia ( CML) Estimating the Efficacy of Nilotinib in Inducing the Persistence of Molecular Remission After Stopping TKI a 2nd or 3rd Time
Brief Title: 2nd or 3rd TKI-stop After 2 Years Nilotinib Pre-treatment in CML-patients
Acronym: NAUT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European LeukemiaNet (Network)
Collaborators: Heidelberg University (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELN-002; 2015-004998-33 (EudraCT Number)
Record Dates: First submitted 2016-03-02; First posted 2016-09-28 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: TKI discontinuation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TKI-stop, pre-treatment with nilotinib (Experimental): Treatment after unsuccessful 1st or 2nd discontinuation at least two year with nilotinib (300 mg/bid). In total, retreatment with TKI for at least 3 years before entering screening for stopping phase is warranted. Clinical monitoring every 3 months during this 2 years.
  Patients who re-achieved and maintained MR4 for at least 12 months and MR4.5 for at least 6 months can enter screening phase for TFR .If MR4.5 is confirmed by an validated laboratory, patient may enter stopping phase of the study. Patient not fulfilling these criteria can be screened again every 3 months until month 48. After TKI-stop hematological monitoring and quantitative PCR of BCR/ABL1 (month 1-6 after stopping: monthly; month 7-12 after stopping: every 1.5 months, thereafter once every three months, for 3 years in total.
  Relapse is defined as BCR-ABL1 > 0.1% on IS at a single time point (loss of MMR) In case of relapse restart of TKI. In general, the same TKI (nilotinib) as before second stop is recommended
  Interventions: Other: TKI discontinuation; Drug: nilotinib

INTERVENTIONS:
Other: TKI discontinuation — 2nd or 3rd TKI stop after pre-treatment with nilotinib.
Drug: nilotinib — Pre-treatment with nilotinib 300 mg/bid for 2 years

SUMMARY:
The main goal of the study is the assessment of duration of major molecular response (MMR) or better at 12 and 36 months after stopping tyrosine kinase inhibitors (TKI) therapy a second or third time in patients with at least three years prior TKI treatment comprising at least two years of nilotinib treatment within this trial and maintained stable MR4 (BCR-ABL ratio <0,01% on international Scale (IS) for at least one year and MR4.5 (BCR-ABL ratio <0,0032% on IS) for at least 6 months:

* who failed a first stop in the EURO-SKI study (standardized criteria)
* who failed a first or second stop outside the EURO-SKI study but would have had fulfilled same eligible criteria and were stopped according to EURO-SKI rules
* who failed a first or second stop outside the EURO-SKI study without fulfilling EURO-SKI rules

DETAILED DESCRIPTION:
The proposal is to re-treat patients with a minimum of two years with nilotinib 2x300 mg/d resulting in total of at least three years TKI treatment who show recurrent disease after unsuccessful first or second stop after TKI treatment in or outside the EURO-SKI study.

If MR4 or better is re-achieved and maintained for at least one year and MR4.5 or better is re-achieved and maintained for at least 6 months, patients will be eligible for a second stop attempt within this study. For MR4, three consecutive PCRs with MR4 or deeper should be measured within one year and for MR4.5, two PCRs during 6 months should demonstrate a MR4.5.

Patients who exhibited hematological relapse after the first stop attempt will not be eligible for a second stop attempt within this study.

After inclusion, 3 monthly monitoring will be performed under nilotinib treatment within the trial. Patients fulfilling the criteria mentioned above will then enter the screening phase.

After verification of MR4.5, TKI treatment will be stopped and patients followed in the same manner as described in EURO-SKI (monthly PCRs for 6 months, 6-weekly PCRs 7-12 months after stopping, thereafter 3-monthly). If MMR is lost (BCR-ABL >0.1% (IS)), TKI treatment will once again be restarted; here the same TKI (nilotinib) is recommended.

It is assumed that after failure of first (or second) stop a switch to treatment with 2GTKI may increase the chance of stopping a second (or third) time [Legros et al. Blood 2012; Rea et al. Blood 2014] It is expected that the rate of a successful second (or third) stop at 12 and 36 months is more than 25%.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with Ph chromosome and/or the BCR-ABL (either b3a2 and /or b2a2) fusion gene positive CML
* CML in CP having failed a prior attempt to stop imatinib or other TKIs therapy either within EURO-SKI or not
* Pretreatment at least one year with any TKI after 1st stop
* Written informed consent

Exclusion Criteria:

* Previous hematological relapse after first stop of TKI.
* Failure to any TKI at any time during CML treatment according to current ELN criteria
* Previous planned or performed allo SCT
* Previous AP/BC at any time in the history of the disease
* High cardiac risk according to ESC score (≥ 10 Points)
* Impaired cardiac function including any of the following:
* Use of a ventricular paced pacemaker; congenital long QT syndrome or family history of; history or presence of significant ventricular or atrial tachyarrhythmias; clinically significant resting bradycardia (<50 bpm); QTcF >450 msec at baseline, myocardial infarction before baseline; other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension).
* Treatment with inhibitors of CYP3A4 or medications that have been well documented to prolong the QT interval is contraindicated.
* History of acute pancreatitis within one year of study entry or medical history of chronic pancreatitis.
* Positive hepatitis B virus serology test or HBV infection
* Any other malignancy except if neither clinically significant nor requires active intervention.
* Severe or uncontrolled medical conditions (i.e., uncontrolled diabetes, acute or chronic liver disease, pancreatic, or severe renal disease unrelated to tumor, active or uncontrolled infection).
* Women who are pregnant, breast feeding, or of childbearing potential without a negative serum pregnancy test at baseline. Male or female patients of childbearing potential unwilling to use an effective barrier contraceptive method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of duration of MMR or better at 12 months after stopping TKI therapy a second or third time | 12 months after stopping
  Assessment of duration of MMR or better at 12 months after stopping TKI therapy a second time in patients with at least three years prior TKI treatment comprising at least two years of nilotinib treatment within this trial and maintained stable MR4 for at least one year and MR4.5 for at least 6 months

SECONDARY OUTCOMES:
Assessment of quality of life (QoL) profiles under nilotinib treatment and comparison with previous TKI therapy before switch and after stopping | 5 years
  To investigate QoL changes over time in relapse-free patients without TKI re-start as measured by the EORTC QLQ-C30 and CML 24 (one combined questionnaire)
Identification of clinical and biological factors correlating with the persistence of MMR or better after stopping TKI | 6 months after stopping
  Proportion of high risk patients according to the risk score at 6 months after stopping TKI;
Estimation of overall survival | 3 years
  Overall survival is calculated from the date of 2nd stop of TKI treatment until the date of death irrespective of the cause of death. Patients still alive at the date of analysis will be censored at the date of last follow-up.
Time to re-achievement of MR4.5 after restart of therapy | 3 years
  Assessment of molecular response after 3 years
Number of patients with grade 1 through grade 5 adverse events (AEs) that are related to study drug, graded according to NCI CTCAE Version 3.0 | 3 years
  Assessment of incidence of any AEs (e.g. from musculoskeletal system) that arise after stopping TKI treatment a second time
Assessment of duration of MMR or better | 36 months after stopping
  Assessment of duration of MMR or better at 36 months after stopping TKI therapy a second or third time in patients with at least three years prior TKI treatment comprising at least two years of nilotinib treatment
Number of patients with grade 1 through grade 5 adverse events (AEs) that are related to study drug, graded according to NCI CTCAE Version 3.0 | 2 years treatment with nilotinib 300 mg/bid
  Assessment of incidence of any AEs (e.g. from musculoskeletal system) that arise after stopping TKI treatment a second time
Estimation of progression-free survival | 3 years
  Progression-free survival is defined as overall survival plus the additional events progression to accelerated phase or blast crisis that also terminate PFS
Identification of clinical and biological factors correlating with the persistence of MMR or better after 6 months | 6 months after stopping
  Proportion of female patients without molecular relapse

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Geiselhart, Study Chair — Heidelberg University
Locations (15):
- Germany (14):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar, München, Bavaria
  - Medizinische Hochschule Hannover, Hannover, North Rhine-Westphalia
  - Universitätsklinikum der RWTH, Aachen
  - Klinikum Bayreuth, Bayreuth
  - Klinikum Chemnitz, Chemnitz
  - Onkologische Schwerpunktpraxis, Esslingen am Neckar
  - Universitätsklinikum Halle (Saale), Halle
  - Schwerpunktpraxis Onkologie, Heilbronn
  - Klinikum der Philipps-Universität, Marburg
  - Kliniken Ostalb, Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Universitätsklinikum Rostock, Rostock
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
- Amsterdam UMC, locatie VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No